CLINICAL TRIAL: NCT07120789
Title: Content, Semantic, and Psychometric Validation of a Patient Knowledge Questionnaire for Pulmonary Hypertension
Brief Title: Validation of a Patient Knowledge Questionnaire for Pulmonary Hypertension
Acronym: SAVOIR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Caio Júlio César dos Santos Fernandes, Principal Investigator, University of Sao Paulo General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: SGP 27073
Record Dates: First submitted 2025-07-04; First posted 2025-08-13 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Pulmonary Arterial Hypertension (PAH); Pulmonary Arterial Hypertension (PAH) (WHO Group 1 PH); Pulmonary Hypertension
Keywords: Pulmonary Hypertension; Patient Knowledge; Questionnaire Validation; Content Validity; Semantic Analysis; Psychometric Validation; Health Education; Patient Education; Chronic Disease
MeSH Terms: conditions — Pulmonary Arterial Hypertension; Hypertension, Pulmonary; Health Education; Chronic Disease

STUDY DESIGN:
Intervention Model Description: This is a methodological study for the development and validation of a questionnaire. The model includes sequential phases: construction, content validation by expert judges, semantic validation with patients, and psychometric analysis in a cross-sectional design. During the final phase, clinical and functional data will be collected from medical records to assess associations between knowledge scores and patient outcomes such as risk stratification (COMPERA 2.0), hospitalizations, and quality of life (CAMPHOR, SF-36, and MBG). The study does not involve any intervention or assignment of participants to treatment arms.
Masking Description: No masking was applied. This is an open-label, non-randomized methodological study to validate a questionnaire. All participants and investigators were aware of the intervention (questionnaire application).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Group (Experimental): Participants in this arm will take part in one of three phases of the questionnaire validation study:
  1. content validation by expert judges,
  2. semantic validation by patients with pulmonary arterial hypertension (PAH),
  3. psychometric validation in a larger sample of up to 200 patients with confirmed PAH.
  In the psychometric phase, participants will complete the final version of the DICTA questionnaire. Additional clinical and functional data will be collected from medical records, including:
  risk stratification using the COMPERA 2.0 method, number of PAH-related hospitalizations, and quality of life scores measured by the CAMPHOR (Cambridge Pulmonary Hypertension Outcome Review), SF-36 (Short Form Health Survey), and MBG (Global Well-Being Measure).
  These data will be used to explore associations between patient knowledge and clinical/functional outcomes.
  Interventions: Other: Application of Patient Knowledge Questionnaire on Pulmonary Hypertension

INTERVENTIONS:
Other: Application of Patient Knowledge Questionnaire on Pulmonary Hypertension — Participants will complete one version of the DICTA questionnaire, developed to assess patient knowledge about pulmonary arterial hypertension. Depending on the study phase, participants will contribute to content validation (expert judges), semantic validation (patients), or psychometric validation (patients). In the final phase, additional data including risk stratification (COMPERA 2.0), hospitalizations, and quality of life scores (CAMPHOR, SF-36, MBG) will be collected for correlational analysis.

SUMMARY:
This methodological study aims to develop and validate a questionnaire named DICTA (Questionnaire for the Assessment of Patient Knowledge in Pulmonary Arterial Hypertension). The study will be conducted in four phases: (1) questionnaire development based on guidelines and literature; (2) content validation by expert judges; (3) semantic validation with patients; and (4) psychometric testing in a sample of up to 200 patients with confirmed pulmonary arterial hypertension (PAH).

In addition to validation, the study will collect clinical and functional data from medical records, including risk stratification using the COMPERA 2.0 method, number of hospitalizations, and quality of life scores assessed by CAMPHOR, SF-36, and MBG. The study will analyze the relationship between patient knowledge (as measured by DICTA) and these outcomes. The final instrument is expected to support patient education strategies and contribute to improved clinical management of PAH.

DETAILED DESCRIPTION:
This is a methodological study with a quantitative approach, developed in four main phases, aimed at constructing and validating a questionnaire to assess the knowledge of patients with pulmonary arterial hypertension (PAH). The study will be conducted at a reference outpatient center in Brazil and will follow established methodological guidelines for the development and validation of health-related instruments.

Phase 1 - Questionnaire Development:

The initial version of the questionnaire, named DICTA, will be created based on the 2022 ESC/ERS Guidelines for PAH, a review of the scientific literature on patient knowledge in chronic diseases, and validated instruments in other conditions (e.g., chronic kidney disease, inflammatory bowel disease, rheumatoid arthritis). Items will cover the following domains: basic concepts, signs and symptoms, diagnosis and exams, available treatments and their mechanisms, adherence and self-care, and side effect management. Items will be multiple-choice with the option "I don't know".

Phase 2 - Content Validation:

At least five expert judges with experience in PAH, health education, and instrument development will evaluate each item for clarity, relevance, representativeness, and appropriateness using a 4-point Likert scale. The Content Validity Index (CVI) will be calculated for each item (I-CVI) and for the total instrument (S-CVI). Items with I-CVI ≥ 0.78 will be retained.

Phase 3 - Semantic Validation:

A sample of at least 10 patients diagnosed with PAH will be asked to complete the questionnaire while verbalizing their understanding ("think-aloud" technique). Revisions will be made based on participant feedback to ensure clarity and comprehension.

Phase 4 - Pilot Study and Psychometric Analysis:

The refined DICTA questionnaire will be applied to a sample of up to 200 patients with confirmed PAH. Psychometric analysis will include internal consistency (Cronbach's alpha) and, if applicable, test-retest reliability (intraclass correlation coefficient - ICC). Exploratory factor analysis may be used to assess internal structure.

In addition to validation, the study will collect clinical and functional data from medical records, including:

Risk stratification using COMPERA 2.0 methodology

Number of hospitalizations related to PAH

Quality of life scores measured by:

CAMPHOR (Cambridge Pulmonary Hypertension Outcome Review)

SF-36 (Short Form Health Survey)

MBG (Medida de Bem-Estar Global)

The relationship between knowledge scores (DICTA) and these outcomes will be analyzed, aiming to explore whether higher patient knowledge is associated with better risk status, lower hospitalization rates, and higher quality of life.

This instrument is expected to help identify educational gaps, support targeted health education strategies, and contribute to improved clinical outcomes and shared decision-making in the care of PAH patients.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older
* Confirmed diagnosis of Group 1 Pulmonary Arterial Hypertension (PAH)
* Ability to read and understand the questionnaire language
* Provided informed consent to participate in the study
* For expert judges (content validation phase): professionals with recognized expertise in pulmonary hypertension, with academic or clinical experience in the field

Exclusion Criteria:

* Cognitive, visual, or auditory impairments that hinder questionnaire comprehension
* Refusal to participate or withdrawal of informed consent
* Inability to complete the questionnaire due to clinical instability

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 215 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Content Validity Index (CVI) of the Questionnaire Items | 4 weeks after expert panel review
  Proportion of agreement among expert judges regarding the relevance and clarity of each item. Items with CVI ≥ 0.80 will be considered valid.
Semantic Clarity Rating by Patients | 2 weeks after patient interview
  Assessment of the clarity and comprehension of each item by patients using a structured form. Items with ≥ 85% of patients rating them as clear or very clear will be considered semantically valid.
Internal Consistency of the Questionnaire (Cronbach's Alpha) | 4 weeks after questionnaire completion
  Psychometric evaluation of the final version of the DICTA questionnaire using Cronbach's alpha. A coefficient ≥ 0.70 will be considered acceptable. The analysis will be conducted in a sample of up to 200 patients.

SECONDARY OUTCOMES:
Test-Retest Reliability (Intraclass Correlation Coefficient - ICC) | 2 weeks after first questionnaire administration
  Stability of the questionnaire scores over time will be assessed by reapplying the instrument after 1 to 2 weeks in a subsample of patients. ICC ≥ 0.80 will be considered acceptable.
Completion Rate and Acceptability of the Questionnaire | At the time of first questionnaire administration (Day 1)
  Percentage of participants who complete the questionnaire without missing data and report that the items are clear and easy to understand.
6. Association Between questionnaire Score and Risk Stratification (COMPERA 2.0) | Within 4 weeks of questionnaire completion
  Association between total DICTA score and patient risk status based on the COMPERA 2.0 stratification tool.
Association Between questionnaire Score and Number of PAH-related Hospitalizations | Within 4 weeks of questionnaire completion
  Correlation between questionnaire score and number of PAH-related hospitalizations in the 12 months prior to questionnaire administration.
Association Between the questionnaire Score (being developed) and Quality of Life Measures (EMPHASIS-10) | Within 4 weeks of questionnaire completion
  Association between questionnaire score and scores on quality of life tools.
Association Between Patient Knowledge and Treatment Adherence using Martin-Bayarre-Grau (MBG Score) | Within 4 weeks of questionnaire completion
  Assess the association between the questionnaire scores and treatment adherence, as measured by the Martin-Bayarre-Grau (MBG) scale. The goal is to explore whether higher knowledge levels are correlated with greater adherence to treatment in patients with pulmonary arterial hypertension.

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto do Coração (InCor), Hospital das Clínicas HCFMUSP, Faculdade de Medicina, Universidade de São Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No